CLINICAL TRIAL: NCT02452671
Title: Observational Plan Designed to Obtain Clinical Experience and Follow up Data on the Use of the ProxiFuse Hammer Toe Device for the Fixation of Osteotomies and Reconstruction of the Lesser Toes Following Correction Procedures
Brief Title: Observational Plan to Obtain Clinical Experience and Follow up Data on the Use of the ProxiFuse Hammer Toe Device
Status: Terminated | Type: Observational
Why Stopped: Enrollment temporarily stopped
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTC-0156
Record Dates: First submitted 2015-05-15; First posted 2015-05-22 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-07

CONDITIONS: Toe Joint Deformity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center, non-randomized, observational study to further evaluate the effectiveness and safety of the Proxifuse Hammer Toe Device when utilized for bone fixation. Approximately 4 US sites will participate. The primary endpoint will evaluate the 6 month post surgery change from baseline in the PROMIS Pain Interference computerized adaptive test (CAT) score.

DETAILED DESCRIPTION:
This is an observational plan designed to obtain clinical experience and follow up data on the use of the ProxiFuse Hammer Toe Device for the fixation of osteotomies and reconstruction of the lesser toes following correction procedures for hammertoe, claw toe and mallet toe.

Collection of data on patients treated with the FDA 510k approved ProxiFuse Hammer Toe Device will assist Cartiva in further evaluation of the effectiveness and safety of the ProxiFuse Hammer Toe Device when utilized for bone fixation per the specified indications. The ProxiFuse Hammer Toe Device is currently approved for commercial distribution and use in the country in which this protocol is being administered (FDA 510k approval K142490). . Given that the product is approved for distribution and use, the product is being used within its approved indication for use, and the data being collected is not burdensome or outside the standard of care, it is determined that no additional regulatory requirements are applicable to this data collection.

The ProxiFuse Hammer Toe Device consists of three components: the implant, deployment instrumentation, and bone awl. The implant is comprised of 2-0 suture, two Nitinol anchors with PEEK Inserts, and a PEEK Stabilizing Body. The device is delivered through a specifically designed instrument. The method of delivery allows for a shifting of the PEEK Body which limits the amount of traction required to place the middle phalanx over the device. The suture utilized in the device serves to shift the PEEK Body and to apply tension between the Nitinol anchors which in turn stabilizes the proximal interphalangeal joint.

In accordance with guidelines as outlined in ISO 14155, ICH GCP, and 21 CFR Part 50, each patient must grant documented informed consent and authorization of disclosure of identifiable health information prior to the collection of clinical data. Each patient should be informed of the procedures to be performed and that data will be collected. It is the intent to use de-identified research data for the potential purposes of product development and publication in marketing literature, journals, and peer-reviewed medical journals.

A copy of the signed informed consent document should be provided to the patient and the original should be maintained as part of the patient's clinical record.

The authorization to use the information collected has no expiration. Cartiva and its affiliates may continue to rely on this authorization to obtain and use the information unless the patient revokes/cancels the authorization in writing. Confidential information will not be shared with anyone outside of Cartiva and its affiliates. Patient names or identifying information will not be used in any reports, publications, or presentations. All data will be de-identified and maintained by University of Rochester .

Data collection will occur at baseline and the following time points after the surgical procedure: 1 week, 6 weeks, 3 months, and 6 months. The study will last for 6 months following each patient's surgical procedures, until the last subject is seen at the 6 month follow up visit, or is withdrawn.

The baseline/preoperative information and assessments should be performed once the subject is consented and enrolled. All operative, discharge, and rehabilitation information should be captured on the eCRFs. Any additional procedures performed during the operation should be documented as well.

The Investigator should complete a foot exam and the subject should complete the PROMIS questionnaires at all clinical follow up visits. The PROMIS data that is collected in this study will be compared to historical AOFAS hammertoe data from the PROMIS database.

Weight bearing anteroposterior and lateral x-rays of the treated toe(s) should be taken at the 1 and 6 week follow up visits. The Investigator should perform a radiographic assessment to observe the presence of any displacements or complications.. Any findings should be captured on the eCRFs.

The following data will be captured on electronic case report forms (eCRFs):

1. Baseline / Preoperative Assessment
2. Operative
3. Follow-up Assessment
4. Adverse Events

CRFs are to be completed by the treating physician or designated clinical representative. Every attempt should be made to provide all CRFs to University of Rochester completed in their entirety for each patient. Where information is not directly available from the patient, a review of the patient's clinical records should be conducted in order to complete as much information as possible on the CRFs.

The sample size for this study is based on the analysis of the primary endpoint. A minimum of 70 patients will be enrolled with the goal of at least 59 patients completing the 6 month visit.

All variables will be analyzed using the intent-to -treat (ITT) data set. The ITT data set will include all enrolled patients who receive the ProxiFuse Hammer Toe device in at least one qualifying toe. No methods will be used to impute values for missing data. Adverse events will be summarized by presenting the number and percent of patients reporting each event.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Has a hammertoe deformity causing daily pain and is a surgical candidate for hammertoe procedure in the 2nd, 3rd and/or 4th toe that has failed non-operative measures
* Capable of completing self-administered questionnaires
* Be willing and able to return for all study-related follow up procedures
* Has not participated in any other research protocol within the last 30 days and will not participate in any other research protocol during this study
* If female, is either using contraception or is postmenopausal, or male partner is using contraception
* Has been informed of the nature of the study, agreeing to its requirements, and have signed the informed consent approved by the IRB

Exclusion Criteria:

* Active bacterial infection of the foot/feet to be treated
* Previous hammertoe correction that requires a revision to a toe to be treated under this study
* Patient is on chronic anticoagulation due to a bleeding disorder or has taken anticoagulants within 10 days prior to surgery
* Muscular imbalance, peripheral vascular disease that prohibits adequate healing, or a poor soft tissue envelope in the surgical field, absence of musculoligamentous supporting structures, or peripheral neuropathy
* Patient is not ambulatory or requires an additional surgical procedure that would prohibit the patient from following standard ProxiFuse post-operative recovery procedures
* Additional foot and ankle surgical procedures required during the index procedure other than foot procedures, lapidus and gastrocnemius recession
* Suspected or known allergic reaction to Nickel or Titanium metals
* Co-morbidity that reduces life expectancy to less than 12 months; or
* Patient is a prisoner or ward of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are candidates for hammer toe surgery.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference computerized adaptive test (CAT) score | Change from baseline at 6 months

SECONDARY OUTCOMES:
PROMIS Pain Interference CAT scores | Change from baseline at 2 weeks; 6 weeks and 3 months after surgery
PROMIS Physical Functioning CAT scores | Change from baseline at 2 weeks; 6 weeks; 3 months and 6 months after surgery
Time to return to normal shoe wear | Time recorded. Subjects will be queried at 2 weeks; 6 weeks; 3 months and 6 months and an actual date recorded. The number of days following surgery will be recorded for analysis
  Normal shoe wear defined as being anything other than a post surgical sandal or boot
Postoperative Adverse Events that require a return to the operating room | From Operative time through 6 months

OTHER OUTCOMES:
PROMIS Pain Intensity short form (SF) | Patient reported outcomes at 2 weeks; 6 weeks ; 3 months and 6 months
PROMIS Depression CAT | Patient reported outcomes at 2 weeks; 6 weeks; 3 months and 6 months
PROMIS Global Health | Patient reported outcomes at 2 weeks; 6 weeks; 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katie Strother, Study Director — Cartiva, Inc.
Locations (5):
- United States (5):
  - Stanford University, Redwood City, California
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan
  - University of Rochester Medical Center, Rochester, New York